CLINICAL TRIAL: NCT03030079
Title: Exploratory Study of Electrical Stimulus as a Treatment Option for Chronic Phantom Limb Pain
Brief Title: Electrical Stimulus Therapy for Chronic Phantom Limb Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Hanger Clinic: Prosthetics & Orthotics (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 16-1063
Record Dates: First submitted 2017-01-13; First posted 2017-01-24 (Estimated); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Phantom Limb Pain
MeSH Terms: conditions — Phantom Limb

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Experimental Electrical stimulation Regimen (Experimental): Explore the efficacy of an electrical stimulus regimen on the treatment of chronic phantom limb pain using a standard-of-care electrical stimulation system
  Interventions: Device: Experimental Electrical Stimulation Regimen

INTERVENTIONS:
Device: Experimental Electrical Stimulation Regimen — The electrodes will pass an electrical current through the skin and into the muscle first at a low intensity for 5 minutes to allow the subject to adjust to the sensation. The current will then be gradually increased to a level sufficient to elicit a non-painful motor contraction. The subject will sit in a relaxed position as the electrical stimulator contracts the muscles for a duration of 15 minutes.
  Other Names: Device: Omnistim FX2 Pro

SUMMARY:
The goal of this pilot study is to assess the effectiveness of an electrical stimulation therapy option for the treatment of chronic phantom limb pain in upper or lower limb amputees. This therapy has been previously used for sports and joint injuries and is marketed for relaxation of muscle spasms, re-education of muscle action, prevention of disuse atrophy, increased local blood circulation, and maintaining or increasing range of motion. The investigators would like to explore the idea that physically exercising the muscles of the residual limb and increasing blood flow to the site of amputation through the promotion of motor contraction using electrical stimulation decreases chronic phantom limb pain.

DETAILED DESCRIPTION:
There are a large number of people living with an amputation due mainly to cardiovascular disease, diabetes, and trauma; and of these there is evidence to show that up to 80% of amputees experience phantom limb pain (PLP). PLP is classified as cramping, burning, shooting, or stabbing pain in the missing limb following an amputation. Current treatments include pharmacological drugs, anesthesia, additional surgery, mirror therapy, transcutaneous electrical nerve stimulation (TENS) and others. TENS, as usually implemented, has been used to effectively reduce pain in multiple spots of the body, but has shown little effect in reducing phantom limb pain especially long term even with varying the frequency and intensity of the electrical stimulation. These current treatments can be invasive, costly, and have shown only to offer immediate relief. Using an electrical stimulator at a higher intensity has proven to to reduce pain and increase healing in numerous sports and joint related injuries. Anecdotally, the investigators have learned that a similar treatment protocol when applied to persons with phantom limb pain can mitigate their pain. The goal of this pilot study is to assess the effectiveness of higher intensity electrical stimulation in the management of PLP and also to acquire data to inform the investigators to the most appropriate study design and power for a future more formal clinical trial. To accomplish this the investigators will utilize the ACP Omnistim FX2 Pro electrical stimulator, that has been provided to us by Accelerated Care Plus (ACP) Corporation, to physically exercise the muscles of the residual limb and hence increase the local blood flow and explore it's potential for treatment of PLP both short and long term. The self-identified subject will be hooked up to the ACP electrical stimulator using surface electrodes that will pass a current through the skin first at a low intensity for 5 minutes to allow the subject to adjust to the tingling sensation. The current will then be gradually increased to a level sufficient to elicit a non-painful motor contraction for 15 minutes. Using a numerical pain scale and short answer questions about the characteristics of the pain the investigators will track both short term and long term changes in pain.

ELIGIBILITY:
Inclusion Criteria:

* Self-identified adult volunteers with a limb deficiency with a well-healed site of amputation
* Subjects experiencing at least a 4 out of 10 of chronic phantom limb pain based on a numeric 10-point pain scale.
* Any ethnicity and gender
* Age (18-85 years)
* Able to understand and follow directions in English, assessed by their ability to respond during the recruitment and consent processes.

Exclusion Criteria:

* Subjects that are not able to understand the procedures and who are unable to come to the facility.
* Any individual whose amputation site is not completely healed
* Anyone with cardiac demand pacemakers and/or implanted defibrillator.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2023-06-27 (Actual); Study Completion 2023-06-28 (Actual)

PRIMARY OUTCOMES:
Use of electrical stimulus medium frequency alternating current for short term decreased Phantom Limb Pan | After each 20 minute treatment session up to 5 weeks
  Pain level data will be taken before and after each session to analyze any short term decreases in pain using a self-reported numeric 10-point pain scale. T- tests will be used for within subject testing looking at pre and post treatment measures to quantify a decrease in pain.
Assess the effectiveness of reducing chronic phantom limb pain long term. | Weekly for 5 weeks
  An overall sustained decrease in phantom limb pain will be assessed weekly using a self-reported numeric 10-point pain scale. ANOVAs will be used to look at trends in post treatment measures over time.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Weir, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- Children's Hospital Colorado Research Institute, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No